CLINICAL TRIAL: NCT00651677
Title: A Multicenter Prospective Randomized Study Comparing Hand Assisted Versus "Pure" Laparoscopic Assisted Proctectomy for Rectal Cancer
Brief Title: Hand Assisted Versus "Pure" Laparoscopic Assisted Proctectomy for Rectal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding issues
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITT02
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2011-04

CONDITIONS: Rectal Cancer
Keywords: hand assisted laparoscopy; rectal cancer; short term outcomes; straight laparoscopy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HAL Proctectomy (Active Comparator): Hand-assisted laparoscopic proctectomy
  Interventions: Procedure: HAL proctectomy; Procedure: Hand-assisted laparoscopic proctectomy
- SL Proctectomy (Active Comparator): "straight" laparoscopic proctectomy
  Interventions: Procedure: "straight" laparoscopic proctectomy; Procedure: SL Proctectomy

INTERVENTIONS:
Procedure: HAL proctectomy — Hand-assisted laparoscopic proctectomy
  Other Names: Gelport
  Arms: HAL Proctectomy
Procedure: "straight" laparoscopic proctectomy — "straight" laparoscopic proctectomy
  Arms: SL Proctectomy
Procedure: Hand-assisted laparoscopic proctectomy — hand-assisted laparoscopic proctectomy
  Other Names: Gelport
  Arms: HAL Proctectomy
Procedure: SL Proctectomy — Straight laparoscopic proctectomy
  Arms: SL Proctectomy

SUMMARY:
We hypothesize that hand-assisted laparoscopy will overcome technical difficulties related to pure laparoscopic rectal surgery and allow surgeons to expand application of laparoscopic techniques to treating patients with rectal cancer. In this study, we plan to randomly assign patients diagnosed with rectal cancer to undergo either "standard" laparoscopic surgery or hand-assisted laparoscopic surgery. We will then compare both peri-operative and long-term outcomes of patients.

DETAILED DESCRIPTION:
Compared to traditional open surgery, laparoscopic surgery for colon cancer results in short-term benefits such as less pain, shorter length of stay, and faster return of bowel function while maintaining equivalent oncologic outcomes. For this reason, increasing numbers of colon cancer patients are undergoing laparoscopic surgery.1-3 Similarly, there are many potential benefits to performing rectal surgery laparoscopically. Although not well documented, laparoscopic rectal surgery is under active study and may result in the usual short-term benefits associated with laparoscopic surgery. In addition, compared to open surgery, laparoscopy can provide unprecedented, unobstructed views of the rectal dissection planes even in a patient with narrow pelvis, not only for the surgeon but to the entire surgical team. Magnified views of the surgical planes allow precise and sharp dissection. The pneumoperitoneum can also help open the planes for mobilization of the mesorectum.

Despite these potential advantages, adoption of laparoscopic rectal surgery has been limited for many reasons. Although there are now several prospective randomized trials demonstrating safety and benefits associated with laparoscopic colon cancer surgery, the same benefits have not yet been clearly demonstrated for laparoscopic rectal cancer surgery.1-3 In addition, concerns about inadequate oncologic rectal dissection, anastomotic complications, and technical challenges have limited wide adaptation of laparoscopic rectal surgery.4,5 In efforts to retain the benefits of laparoscopic surgery while not compromising oncologic rectal dissection, others have advocated performing hybrid procedures in which colonic portion of the surgery is performed using the "pure" laparoscopic technique and rectal dissection is performed open through a limited low midline or Pfannestiel (low transverse) incision.6

Hand-assisted laparoscopic surgery is a technique in which the surgeon places a hand into the abdomen through an airtight access device while performing laparoscopic surgery. By placing a hand into the abdomen during laparoscopy, surgeons retain their abilities to manually retract, expose, and manually dissect, which are lost in pure laparoscopic surgery. Retention of these abilities can significantly expedite the operation. In fact, several studies have demonstrated that hand-assisted laparoscopic colon surgery results in significantly shorter operative time and less conversion to open surgery while maintain similar short-term outcomes compared to "pure" laparoscopic technique.7-9 In rectal surgery for cancer, sigmoid colon, left colon, and splenic flexure need to be mobilized in order to allow tension free anastomosis between the colon and the residual rectum. In laparoscopic proctectomy, HALS compared to SLS technique may therefore, result in shorter operative time based on colonic portion of the operation alone.

One of the technical hurdles in performing laparoscopic rectal dissection is exposure and retraction of the rectum. As one dissects down to the distal rectum, especially in patients with narrow pelvis, crowding and clashing of instruments can result in poor exposure and dissection. The only prospective randomized trial comparing results of open vs. laparoscopic surgery to include rectal cancer is CLASICC trial.3 It reported an increased circumferentially positive margin of cancer following laparoscopic rectal resection with twice as many patients in the laparoscopic group (12 %) having an involved margin as in the open group (6 %). This increased radial margin may be related to difficulty in retraction and exposure. In HALS, rectal exposure and dissection can be either performed directly through the incision using the open techniques or laparoscopically with manual assistance. This may result in equivalent oncologic outcomes as the open surgery but with shorter operative time compared to SLS technique.

A further challenge in laparoscopic rectal surgery is localization of the tumor, which is less of an issue in colon cancer where the tumor is easily visible or tattooed preoperatively. This is not possible for rectal cancer, which can pose a problem in both dissection and safe division of the rectum. Without tactile sensation it can be difficult to be sure that the stapler is below the tumor. Hand assisted laparoscopic surgery allows preservation of tactile sensation and therefore circumvent the above problem. The next step following mobilization of the rectum is division of the rectum and anastomosis. This poses a challenge for the laparoscopic surgeon for several reasons. The current laparoscopic stapling devices angulate to a maximum of 65 o making horizontal division of the rectum difficult. Morin et al reported a leak rate of 17 % below 12 cm from the anal verge and as high as 25 % in those who were not diverted following laparoscopic rectal surgery.4 Leroy et al reported a similar leak rate of 20 % in cancers below 15 cm following laparoscopic rectal surgery.5 Comparatively higher leak rates after laparoscopic rectal surgery may be related to limitations in currently available laparoscopic surgical staplers. By performing distal rectal division through the incision by using the open surgical staplers, hand-assisted laparoscopic rectal surgery may result in lower anastomotic leakage rate.

We hypothesize that hand-assisted laparoscopy may result in shorter operative time while retaining the benefits associated with laparoscopic surgery. In this study, we plan to randomly assign patients diagnosed with rectal cancer to undergo either "standard" laparoscopic surgery or hand-assisted laparoscopic surgery. We will then compare both peri-operative and long-term outcomes of patients. If our hypothesis is true, hand assisted laparoscopic approach to rectal surgery may be preferable to standard laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > = 18 years of age
* Histologically proven rectal cancer
* Inferior margin of the cancer located within 15 cm from the anal verge as determined by rigid sigmoidoscopy
* No evidence of distant metastases
* Childbearing age women with negative pregnancy test
* Patient is a candidate for elective rectal resection
* The patient, or their representative, is able to understand the study and is willing to consent to participation in the study.

Exclusion Criteria:

* Age < 18 years of age
* Surgically unresectable rectal cancer
* Patients who will require APR or hand-sewn colo-anal anastomosis
* ASA class 4 or 5
* Patients having additional surgical procedures which may have affect recovery
* Child bearing age women with positive pregnancy test
* Patients with contraindication for treatment by laparoscopy
* Patients or their representative who are unable to understand the conditions and objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
operative time | post-operative

SECONDARY OUTCOMES:
Adequacy of resection margins | post-operative
In-hospital mortality and morbidity | during hospitalization
urinary and sexual function | preoperative and 3-6 months postop

CONTACTS AND LOCATIONS:
Overall Officials: Sang W Lee, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Sang Lee, New York, New York, United States